CLINICAL TRIAL: NCT04828109
Title: A Digital Intervention Protocol to Enhance Recovery After Head and Neck Surgery
Brief Title: Digital Intervention Postoperative Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00021902
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Surgery; Otolaryngologic Disorder; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR and Fitbit (Active Comparator): Daily VR use every 3 hours up to 30 minutes at a time and Fitbit daily step goal of 2,000 steps
  Interventions: Device: Virtual Reality; Device: Fitbit
- VR Only (Active Comparator): Daily VR only. Daily VR use every 3 hours up to 30 minutes at a time.
  Interventions: Device: Virtual Reality
- Fitbit Only (Active Comparator): Fitbit daily step goal of 2,000 steps.
  Interventions: Device: Fitbit
- Control (No Intervention): Standard of care

INTERVENTIONS:
Device: Virtual Reality — Use of any virtual reality experiences available
  Arms: VR Only; VR and Fitbit
Device: Fitbit — Use of a Fitbit wearable activity device to track daily step goals.
  Arms: Fitbit Only; VR and Fitbit

SUMMARY:
Postoperative recovery after head and neck surgery is complex, and often requires utilization of narcotic medications. The aim of this study is to evaluate reduction in pain and use of opioid medications through Virtual Reality (VR) and Fitbit wearable activity devices.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) protocols were introduced as a method to optimize perioperative patient care. Narcotic medications are frequently utilized in postoperative care, but these have risks including sedation or dependence. Non-pharmacologic measures for postoperative pain control may help limit the need for opioids in postoperative pain control.

Early mobilization is also important after surgery, however postoperative mobility is rarely monitored and relies on subjective reports.

The investigators will seek to examine the implementation of an ERAS protocol using VR and Fitbit wearable activity devices on postoperative recovery after head and neck surgery. This is a prospective, 4-arm, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18 to 89 years of age.
* Planned to undergo major head and neck surgery OHSU with an expected length of stay of two days or more.
* Ability to understand goals of the study and willingness to sign a written informed consent document.

Exclusion Criteria:

* Planned postoperative admission to the intensive care unit (ICU).
* Social or psychiatric conditions that may interfere with compliance.
* Isolation precautions.
* Reconstruction, incisions, wounds, wound care, or injury that impact the ability to place on the VR headset or wear a Fitbit device around the wrist.
* History of seizure or epilepsy.
* History of vertigo or persistent dizziness.
* Limitations that impair mobility.
* Use of a walker or wheelchair at baseline.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Mean daily opioid use | through study completion, an average of 10 days
  Mean daily opioid use will be assessed converted into milligram morphine equivalents (MME).

SECONDARY OUTCOMES:
Pain scores | through study completion, an average of 10 days
  The Numeric Rating Scale (NRS) from 0 to 10 will be used to determine pain scores collected in the morning and evening each day. Scores will be averaged to obtain the daily pain score. We will also look at differences between AM and PM pain scores among the different cohorts. Scores will range from 0 (no pain) to 10 (worst pain)
Anxiety | Before surgery and at study completion, an average of 10 days
  The Generalized Anxiety Disorder 7-Item scale (GAD-7) will be used to determine preoperative and postoperative level of anxiety. Cut points of 5, 10, and 15 may represent mild, moderate, and severe levels of anxiety.
Depression | Before surgery and at study completion, an average of 10 days
  The Patient Health Questionaire-9 (PHQ-9) will be used to determine preoperative and postoperative level of depression. PHQ-9 scores can represent mild (<4), moderate (5-14), and severe (>20) depression.
Sleep Quality | Before surgery and at study completion, an average of 10 days
  The Insomnia Severity Index (ISI) will be used to determine preoperative and postoperative sleep quality. The ISI is a 7-item questionnaire evaluating severity of difficulty with sleep onset, sleep maintenance, early morning awakening, sleep dissatisfaction, interference in daytime functioning, noticeability of sleep difficulties by others, and distress from sleep difficulty. Items are rated on a 5-point Likert scale, and a total score ranges from 0 to 28.
Patient experience and satisfaction | at study completion, an average of 10 days
  A Visual Analogue Scale (VAS) will used to analyze patient satisfaction during hospitalization, and will be provided to patients on day of discharge. The VAS is a horizontal line that is 100-mm long, with no satisfaction (0) on the very left and extreme satisfaction on the very right (100).
Disposition on discharge | at study completion, an average of 10 days
  Data regarding disposition on discharge to home, home with home health, skilled nursing facility, inpatient rehabilitation facility, or other facility will be determined from the electronic medical record on the day of discharge.
Length of hospital stay | at study completion, an average of 10 days
  Length of stay will be calculated beginning from postoperative day one and will include the day of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Li, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No